CLINICAL TRIAL: NCT00713206
Title: A Prospective, Randomized-Controlled, Multicenter Study of NanoTite Implants Placed Into Fresh Sinus Lift Augmentation Sites
Brief Title: Prospective Study of NanoTite Implants Placed Into Fresh Sinus-Lift Augmentation Sites (VSSL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2604
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Tooth Disease; Partial Edentulism
Keywords: Dental implants, maxilla, sinus lift, augmentation
MeSH Terms: conditions — Tooth Diseases | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dental implant (Osseotite) (Active Comparator): Dental implants placed simultaneously with graft augmentation material.
  Interventions: Device: Dental Implant (Osseotite)
- Control group (No Intervention): Dental implants placed into graft augmentation material that has four months to heal.

INTERVENTIONS:
Device: Dental Implant (Osseotite) — Root form titanium dental implant
  Other Names: Osseotite
  Arms: Dental implant (Osseotite)

SUMMARY:
This prospective, randomized-controlled, clinical study evaluates the ability of the NanoTite implant system to achieve integration and provide long-term support of a prosthesis when placed immediately in fresh sinus augmentation material. Control cases will be those where the sinus augmentation material is allowed four months of healing prior to NanoTite implant placement. In addition to implant performance, radiographic evidence of crestal bone regressive modeling will be used to evaluate differences between test and control cases.

Study (null) hypothesis: The implants placed into sinus augmentation sites at the time of grafting will have the same integration success and maintenance of integration as for the implants placed after four months of graft healing.

DETAILED DESCRIPTION:
This will be a prospective, randomized-controlled, longitudinal study in which qualified patients with partial edentulism and thin maxillary ridges will have as part of their treatment at least one sinus ridge augmentation procedure and have their edentulism restored with an implant-supported short-span or long-span fixed bridge. Each patient may have up to two cases included in the study should they need bilateral sinus augmentation using unilateral bridge restorations on either side.

Each patient (or side if a bilateral case) will be randomly assigned to one of two groups: Treatment Group 1 (test) cases will have implants placed into the sinus cavity during the graft augmentation procedure. Treatment Group 2 (control) will have a sinus lift augmentation and implant placement into this area will take place after four months of graft healing. For both groups the implants will be submerged and allowed four months of healing before second stage surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and any race greater than 18 years of age
* Patients for whom a decision has already been made to augment one or both maxillary sinuses for the purpose of placing dental implants in a maxillary ridge no less than 3 mm high and no greater than 5 mm in height
* Patients must be physically able to tolerate conventional surgical and restorative procedures.
* Patients must agree to be evaluated for each study visit, especially the yearly follow-up visit

Exclusion Criteria:

* Patients with active infection or severe inflammation in the areas intended for implant placement.
* Patients with a >10 cigarettes per day smoking habit.
* Patients with uncontrolled diabetes mellitus.
* Treatment with therapeutic radiation to the head within the past 12 months.
* Patients who are pregnant at the screening visit.
* Patients with evidence of severe para-functional habits such as bruxing or clenching.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Caputi, DDS, Principal Investigator — Director del Dipartimento di Scienze Odontostomatologiche
Locations (1):
- Università "G. d' Annunzio" Chieti-Pescara, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in the study according to inclusion/ exclusion criteria as described in the protocol. Patient enrollment began September 2006 and ended May 2008.
Units Other Than Participants: dental implant
Groups:
- Treatment Group: Dental implants placed simultaneously with graft augmentation material.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 65; 158 dental implant | 57; 140 dental implant
Completed | 60; 152 dental implant | 53; 131 dental implant
Not Completed | 5; 6 dental implant | 4; 9 dental implant
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 62 | 30 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 23 | 83
  >=65 years | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 17 | 45
  Male | 34 | 13 | 47
Region of Enrollment [Number; unit: participants]
  Italy | 44 | 19 | 63
  Spain | 9 | 5 | 14
  Portugal | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Implants Not Mobile (Not Failing) at End of 3 Years
Description: All surviving implants at the end of study (3 years)
Time Frame: 3 years
Population: dental implants
Measure: Number; unit: dental implant
Units Other Than Participants: dental implant
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 65 | 57
Number analyzed (dental implant) | 158 | 140
dental implant | 158 | 140

2. Other Pre Specified Outcome: Crestal Bone Loss (Measured Value of Bone Level Around the Dental Implant)
Description: Average measured bone loss (change from baseline) for each implant placed at 3 years final time frame
Time Frame: 3 year
Reporting Status: Not Posted, anticipated posting 2024-07

ADVERSE EVENTS:
Time Frame: Adverse events are collected and reported from day 1 up to 3 years (end of the study)
Description: Adverse event data is collected by patient questioning and visual examination of patient's mouth during each study visit
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/57
Other Adverse Events (participants affected / at risk) | 2/65 | 1/57
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=65) | Control Group (N=57)
Mobility (Surgical and medical procedures) | 2 (65) | 1 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.